CLINICAL TRIAL: NCT04869384
Title: Effect of Electronic Monitoring and Feedback on Adherence to Easyhaler Controller Medication in Patients With Asthma
Acronym: eMOFEE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3103017; 2019-003082-17 (EudraCT Number)
Record Dates: First submitted 2021-04-27; First posted 2021-05-03 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Subjects will receive reminders and feedback to improve their adherence via a sensor attached to Easyhaler inhaler and mobile application
  Interventions: Other: Reminders and feedback to improve adherence
- Usual care (Active Comparator): Subjects do not receive reminders and feedback, but receive treatment as usual.
  Interventions: Other: No reminders and feedback to improve adherence

INTERVENTIONS:
Other: Reminders and feedback to improve adherence — Subjects will receive reminders and feedback to improve their adherence.
  Arms: Intervention
Other: No reminders and feedback to improve adherence — Subjects will not receive reminders and feedback to improve their adherence.
  Arms: Usual care

SUMMARY:
Effect of Electronic Monitoring and Feedback on Adherence to Easyhaler Controller Medication in Patients with Asthma

ELIGIBILITY:
Main inclusion Criteria:

* written informed consent
* male and female subjects with documented diagnosis of asthma
* age 18 to 65 years
* ACT score 19 or less at screening
* treatment wih oral corticosteroids or hospital or emergency department admission due to asthma exacerbation within the past year
* subject's able to use Easyhaler inhalers and comply with study requirements

Main exclusion Criteria:

* recent (within 1 month) asthma exacerbation
* concomitant major respiratory disease which may complicate the measurement of asthma control
* >20 pack-year history of smoking
* recent upper or lower respiratory tract infection
* pregnant or lactating female subjects

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2021-06-23 (Actual); Primary Completion 2024-04-24 (Actual); Study Completion 2024-04-24 (Actual)

PRIMARY OUTCOMES:
Mean weekly adherence to controller medication | Weekly during each of the last 6 weeks of treatment
  Adherence (percentage of doses taken of the doses prescribed) to controller medication during last six weeks of study

CONTACTS AND LOCATIONS:
Overall Officials: Orion Corporation Clinical Study Director, Study Director — Orion Corporation, Orion Pharma
Locations (1):
- MECS Research GmbH, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No